CLINICAL TRIAL: NCT05749133
Title: An Investigator-initiated Trial Evaluating the Efficacy and Safety of Anti-GPRC5D CAR-T Cells Therapy in Patients With Relapsed / Refractory(r/r) Multiple Myeloma(MM) Who Have Received Third-line or More Treatments
Brief Title: Safety and Efficacy of Anti-GPRC5D CAR-T Cells Therapy in the Treatment of r/r MM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: XuYan (Other)
Responsible Party: Sponsor-Investigator, XuYan, Associate chief physician, Institute of Hematology & Blood Diseases Hospital, China
Organization: Institute of Hematology & Blood Diseases Hospital, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG-CT-22-011
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma, Refractory
Keywords: CAR-T
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-GPRC5D CAR-T (Experimental): Subjects who meet the enrollment conditions will receive intravenous infusion of Anti-GPRC5D CAR-T Cells Injection, doses of 1.0~6.0×10^6 /kg±20% CAR-T cells, after lymphodepleting therapy.
  Interventions: Biological: Anti-GPRC5D CAR-T Cells Injection

INTERVENTIONS:
Biological: Anti-GPRC5D CAR-T Cells Injection — This is a"3+3"dose escalation study, in which three dose groups are set three different dose levels of CAR-T cells: Initial dose group: 3.0×10^6/kg±20%; Low dose group: 3.0×10^6/kg±20%; High dose group: 6.0×10^6/kg±20%. Dose was weight-based.

SUMMARY:
It is a single-center, open-labeled, single-arm, non-randomized investigatorinitiated trial evaluating the efficacy and safety of anti-GPRC5D CAR-T cells therapy for relapsed and refractory(r/r) multiple myeloma(MM) after three or more lines of treatments.

DETAILED DESCRIPTION:
This open label, single-arm, investigator-initiated study aims to evaluate the efficacy and safety of Anti-GPRC5D CAR-T in subjects with relapsed and refractory(r/r) multiple myeloma(MM) after three or more lines of treatments. A leukapheresis procedure will be performed to manufacture Anti-GPRC5D chimeric antigen receptor (CAR) modified T cells. Prior to Anti-GPRC5D CAR-T cells infusion subjects will receive lymphodepleting therapy with fludarabine and cyclophosphamide. After infusion, the safety and efficacy of CAR-T therapy was evaluated by investigators.

ELIGIBILITY:
Inclusion Criteria:

1. The patient understands and voluntarily signs the informed consent, and is expected to complete the follow-up examination and treatment of the study procedure.
2. Age 18 to 75 years old, gender is not limited.
3. Diagnosed with multiple myeloma according to IMWG diagnostic criteria.
4. Have received third-line or above treatment.
5. Have measurable lesions at screening period, defined as any of the following : (1) serum monoclonal immunoglobulin (M-protein) level ≥1.0 g/dL. (2) urine M protein level ≥200 mg/ 24h. (3) Light chain multiple myeloma diagnosed with no measurable lesion in serum or urine: serum immunoglobulin free light chain is ≥10 mg/dL and serum immunoglobulin κ/γ free light chain ratio is abnormal.
6. The patient has recovered from the toxicity of the previous treatment, that is, the CTCAE toxicity grade is less than 2 (unless the abnormality is related to the tumor or is in a stable state as judged by the investigator, which has little effect on safety or efficacy).
7. Eastern cooperative oncology group (ECOG) score is 0-2, and survival is expected to be greater than 3 months.
8. Has proper organ function: (1) Alanine aminotransferase (ALT) ≤3 times the upper limit of normal (ULN). (2) Aspartate aminotransferase (AST) ≤3 times ULN. (3) Total bilirubin ≤1.5 ULN. (4) Serum creatinine ≤1.5 ULN, or creatinine clearance ≥60 mL/min. (5) Indoor oxygen saturation ≥92%. (6) Left ventricular ejection fraction (LVEF) ≥45%, echocardiography confirmed no pericardial effusion, no ECG findings with clinical sense. (6) There was no clinically significant pleural effusion.
9. The venous access required for collection can be established, and there are no contraindications to leukocyte collection.

Exclusion Criteria:

1. Have been diagnosed with or treated for aggressive malignancies other than multiple myeloma within 3 years.
2. Subjects who have received the following therapies before blood collection: have received targeted therapy, epigenetic therapy, or investigational drug therapy or invasive investigational medical device within 14 days or at least five half-lives, whichever is shorter, or have treated with monoclonal antibodies within 21 days, or have received cytotoxic therapy within 14 days, or have treated with a proteasome inhibitor within 14 days, or have treated with an immunomodulatory agent within 7 days, or have received radiotherapy within 14 days (except bone marrow reserve with field coverage ≤ 5%).
3. It is suspected that MM has involved the central nervous system or meninges and has been confirmed by MRI or CT, or there are other active central nervous system diseases.
4. Patients with macroglobulinemia, POEMS syndrome (polyneuropathy, organ enlargement, endocrine disease, monoclonal proteinosis, and skin changes) or primary AL amyloidosis at the time of screening.
5. Hepatitis B surface antigen (HBsAg) is positive, or Hepatitis B core antibody (HBcAb) positive while HBV DNA titer in peripheral blood higher than the lower limit of detection. Hepatitis C virus (HCV) antibody positive and the peripheral blood HCV RNA also positive. Human immunodeficiency virus (HIV) antibody positive. Cytomegalovirus (CMV) DNA test results ≥500 copies /mL. Syphilis test positive.
6. Those with a history of severe allergies or known any of the active ingredients, excipients or mouse-derived products contained in the drug, or those allergic to xenogeneic proteins in this trial, including lymphocyte depletion regimens. Severe allergy history is defined as an allergic reaction of grade two or above, and any of the following clinical manifestations occur when an allergic reaction occurs: airway obstruction (runny nose, cough, wheezing, dyspnea), hypercardia tachycardia, hypotension, arrhythmia, gastrointestinal symptoms (nausea, vomiting), incontinence, laryngeal edema, bronchospasm, cyanosis, shock, respiration, cardiac arrest.
7. Severe heart disease, including but not limited to severe arrhythmia, unstable angina, massive myocardial infarction, New York Heart Association class III or IV cardiac insufficiency, refractory hypertension (refractory Hypertension is defined as: on the basis of improving lifestyle, a reasonable tolerable and sufficient amount of ≥3 kinds of antihypertensive drugs (including diuretics) has been used for > 1 month and the blood pressure has not reached the standard, or the blood pressure can only be achieved effective control after taking ≥4 kinds of antihypertensive drugs.
8. Systemic diseases judged by investigators to be unstable, including but not limited to severe liver, kidney or metabolic diseases requiring drug treatment.
9. Patients with acute/chronic graft-versus-host disease (GVHD) within 6 months prior to screening, or requiring immunosuppressive therapy for GVHD.
10. Active autoimmune or inflammatory diseases of the nervous system (eg, Guillain-Barre syndrome (GBS), amyotrophic lateral sclerosis (ALS)) and clinically significant active cerebrovascular disease (eg, cerebral edema) , Posterior Reversible Encephalopathy Syndrome (PRES)).
11. Those who have tumor emergencies (such as spinal cord compression, intestinal obstruction, leukostasis, tumor lysis syndrome, etc.) before screening or reinfusion and need emergency treatment.
12. The presence of an uncontrolled bacterial, fungal, viral or other infection requiring antibiotic treatment.
13. Those who have undergone major surgical operations (except diagnostic surgery and biopsy) within 4 weeks before clearing the lymph cells, or those who plan to undergo major surgery during the study period, or those whose surgical wounds have not healed completely before enrollment.
14. Those who have received (attenuated) live virus vaccine within 4 weeks before screening.
15. Persons with severe mental illness.
16. Those who are alcoholics or have a history of drug abuse.
17. Pregnant or lactating women, female subjects who plan to have a pregnancy within 2 years after cell infusion, and male subjects whose partners plan to have a pregnancy within 2 years after cell infusion.
18. Patients who are contraindicated with any study procedure or have other medical conditions that may expose them to unacceptable risks in accordance with the investigator's judgment and/or clinical standards. 19. Patients who, in the judgment of the investigator and/or clinical standards, are contraindicated with any study procedure or have other medical conditions that may expose them to unacceptable risks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events(AE) after infusion | Up to the subject withdrew or 24 months after CAR-T infusion.
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included. Description, time, classification, and outcome of AE events resulted from the investigational medical product, delivery method, or emergency measures will be recorded in the case report form.
Dose limited toxicity (DLT) | Up to 28 days after infusion.
  Dose limited toxicity(DLT) was defined as the occurrence of any of the following adverse events within 28 days of the infusion of CAR-T cells after optimal supportive treatment, which were discussed with the investigator and determined to be associated or likely to be associated with the infusion.
Overall response rate(ORR) | Day 28 and months 3, 6, 9, 12, 18, 24 after CAR-T infusion.
  Overall Response Rate (ORR) is defined as the proportion of subjects achieving strict complete remission(sCR), complete response(CR), very good partial response(VGPR) and partial response(PR).
Clinical benefit rate | Day 28 and months 3, 6, 9, 12, 18, 24 after CAR-T infusion.
  It's defined as the sum of the proportion of subjects who achieved ORR (sCR + CR + VGPR + PR) and minimal response (MR) according to the International Myeloma Working Group (IMWG) criteria.
Progression-free survival(PFS) | Up to 24 months after CAR-T infusion.
  Progression-free survival(PFS) refers to the time from cell reinfusion to the first assessment of tumor progression or death from any cause.
Overall survival(OS) | Up to 24 months after CAR-T infusion.
  Overall survival (OS) refers to the time from the time the patient received an infusion of CAR-T cells until death (from any cause).

SECONDARY OUTCOMES:
Concentration of CAR-T cells | Up to 3 months after CAR-T infusion.
  Concentration of CAR-T cells measured by Flow cytometry after CAR-T infusion.
Concentration of cytokine | Up to 28 days after CAR-T infusion.
  Concentration of CAR-T cells measured by ELISA or other methods after CAR-T infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Xu, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China